CLINICAL TRIAL: NCT05839730
Title: Fast Induced Remodeling in Heart Failure With Preserved Ejection Fraction
Acronym: FIRE-HFpEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: MDT20060
Record Dates: First submitted 2023-03-01; First posted 2023-05-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Concentric Hypertrophy

STUDY DESIGN:
Intervention Model Description: Eligible subjects will have enrollment data collected, including a blood draw. Subjects will then have a pacemaker implanted. After 6 weeks, subjects will have a follow up visit with a blood draw and a cardiac MRI. At this visit, subjects will be randomized 2:1 for pacing therapy or as a control (programmed into either a non-pacing mode or an exertional rate-adaptive pacing mode with no planned pacing at rest). After 3, 6 and 9 months after randomization, subjects will return for a follow up visit. At the 9-month visit therapy modifications will be made based on initial pacing randomization assignment: pacing therapy will be terminated in the original therapy group and enabled in the control group. After an additional 3-months of follow-up, subjects will return for their final visit, therapies will be disabled in all subjects and subjects will be exited.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects and assessors of outcomes will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Pacemaker with multiple pacing therapies enabled (Experimental): Device will be programmed for personalized lower rate pacing (PLR) and tachycardiac remodeling pacing (TRT).
  Interventions: Device: Pacemaker PLR + TRT ON
- Pacemaker with no pacing therapies enabled (Active Comparator): Device will be programmed to a non-pacing mode or an exertional rate-adaptive pacing mode with no planned pacing at rest.
  Interventions: Device: Pacemaker non-pacing mode or an exertional rate-adaptive pacing mode with no planned pacing at rest.

INTERVENTIONS:
Device: Pacemaker PLR + TRT ON — RAMware modified implantable pulse generator (IPG) with personalized lower rate (PLR) and tachycardia remodeling therapy (TRT) ON
  Arms: Pacemaker with multiple pacing therapies enabled
Device: Pacemaker non-pacing mode or an exertional rate-adaptive pacing mode with no planned pacing at rest. — RAMware modified implantable pulse generator (IPG)
  Arms: Pacemaker with no pacing therapies enabled

SUMMARY:
FIRE-HFpEF is a multi-center, prospective, randomized, single-blinded, clinical feasibility study. This study will enroll up to 105 subjects with heart failure with preserved ejection fraction in the United States. Data will be collected to evaluate whether pacing therapies can lead to improvements in exercise capacity and health status of subjects.

DETAILED DESCRIPTION:
After enrollment, baseline data will be collected, and subjects will then have a pacemaker implanted. After 6 weeks, subjects will have a follow up visit with a blood draw and a cardiac MRI. At this visit, subjects will be randomized 2:1 for pacing therapy or as a control (programmed into either a non-pacing mode or an exertional rate-adaptive pacing mode with no planned pacing at rest). After 3, 6 and 9 months after randomization, subjects will return for a follow up visit. At the 9-month visit therapy modifications will be made based on initial pacing randomization assignment: pacing therapy will be terminated in the original therapy group and enabled in the control group. After an additional 3-months of follow-up, subjects will return for their final visit, therapies will be disabled in all subjects and subjects will be exited. Echocardiographic, functional, and health status endpoints will be collected and analyzed to assess therapy efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Heart Failure, Left Ventricular Ejection Fraction (LVEF) ≥ 55% (this and other measurements must be made within the last year).
* New York Heart Association (NYHA) Functional Class I-III
* Stable on guideline-directed medical therapy (GDMT) heart failure medications as determined by the investigator, for at least 1 month, with the exception of loop diuretic therapy. GDMT should be in accordance with current American Heart Association (AHA)/American College of Cardiology (ACC)/Heart Failure Society of America (HFSA) Guidelines and include consideration of Sodium/glucose cotransporter-2 inhibitors (SGLT2i) therapy.
* V End Diastolic Volume indexed to body surface area (BSA) ≤ 80 mL/m^2.
* Concentric remodeling or concentric hypertrophy defined as at least one of the following criteria:

  * Left ventricular (LV) posterior or lateral wall thickness > 11mm
  * Relative wall thickness (RWT) > 0.42
  * Male and LV mass indexed to BSA ≥115 g/m2
  * Male and LV mass indexed to height ≥ 49.2 g/m2.7
  * Female and LV mass indexed to BSA ≥ 95 g/m2
  * Female and LV mass indexed to height ≥ 46.7 g/m2.7

Exclusion Criteria:

* Unable or unwilling to undergo contrast MRI.
* Class I indication for permanent pacing, except for symptomatic chronotropic incompetence
* Current permanent or persistent Atrial fibrillation (A-fib)
* Structural heart disease requiring intervention
* Aortic valve replacement procedure less than 12 months prior to enrollment
* Known pericardial constriction, genetic hypertrophic cardiomyopathy, or infiltrative cardiomyopathy
* Severe aortic or mitral valve disease, defined as severe regurgitation or a valve area < 1cm^2
* Exertional angina
* Severe pulmonary disease including severe Chronic obstructive pulmonary disease (COPD) (i.e., requiring home oxygen, chronic nebulizer therapy, or chronic oral steroid therapy or hospitalized for pulmonary decompensation within 12 months)
* Estimated glomerular filtration rate (eGFR) < 25 ml/min/1.73m^2 as calculated by the Modification in Diet in Renal Disease (MDRD) formula
* Uncontrolled blood pressure, defined as systolic pressure outside the range of 100 to 160 mmHg despite anti-hypertensive medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
characterize the effect of TRT + PLR on cardiac structure. LV mass, LVEDV, LVESV, and wall thickness which will be collected at baseline, 3-month, 6-month, 9-month, and 12-month visits. | Through study completion, projected for three years until last subject last 12-month visit.
Characterize the effect of pacing therapies on health status, defined as change in the Minnesota Living with Heart Failure Questionnaire (MLHFQ) from baseline to 3, 6, and 9 months. | Through study completion, projected for three years until last subject last 12-month visit.
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) is a validated patient-oriented measure of the adverse effects of heart failure on a patient's life. Each of the 21 questions are scored on a 6-point Likert Scale (0 to 5), the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life.
Characterize the durability of cardiac remodeling changes and assess the safety and tolerability of TRT + PLR. | Through study completion, projected for three years until last subject last 12-month visit.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - NCH Heart Institute, Naples, Florida
  - Prairie Education and Research Cooperative-St. Elizabeth's, O'Fallon, Illinois
  - Prairie Education and Research Cooperative-St. John's, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Duke University, Durham, North Carolina
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Dallas VA Medical Center, Dallas, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - The University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No